CLINICAL TRIAL: NCT05440994
Title: Phenotypic Description of Patients With Atypical Clinical Forms of PLA2G6 Mutations
Acronym: ATYPICPLA2G6
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2021 SARRET ATYPIC-PLA2G6
Record Dates: First submitted 2022-06-07; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-05

CONDITIONS: Neuroaxonal Dystrophy, Atypical
Keywords: PLA2G6; atypical infantile neuro-axonal dystrophy; progressive ataxia; Karak syndrome; pediatric parkinsonism; cerebello-spastic syndrome
MeSH Terms: conditions — NBIA2B; Karak Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mutations in the PLA2G6 gene are well known in the classical phenotype called infantile neuro-axonal dystrophy (INAD), a severe neurodegenerative disease starting in infancy with homogeneous clinical, radiological, electrophysiological and pathophysiological features, with early death. Other clinical forms in pediatric patients called atypic INAD have been described in some patients. Expansion of high-throughput sequencing in the last decades has lead to identify mutations in the PLA2G6 gene in pediatric patients with late-onset phenotypes associating progressive ataxia, spastic paraplegia, cognitive regression and/or dystonia / parkinsonism. A high variability in radiological and electrophysiological findings is also described. Less than twenty patients with a pediatric onset have been reported with an atypical INAD. Very poor data are available on management and therapeutic options in these patients and global prognostic is not known. This multicentric retrospective study will record clinical, radiological, electrophysiological and pathophysiological data in pediatric patients with genetically confirmed atypical INAD. Management, therapeutics and evolution of the disease will also be recorded.

DETAILED DESCRIPTION:
Patients with biallelic mutations in PLA2G6 with an atypic INAD starting before 18 years will be recruited after a collaboration call of neuropaediatricians in France. After family consent, a retrospective collection of data will be performed using REDCap® digital questionnaire performed by the practitioner who follows / followed each patient.

Genetical, clinical, radiological, electrophysiological, pathophysiological outcomes will be anonymously recorded. Therapeutics proposed to patients, potential complications of the disease or treatments, age of premature death will also be recorded.

Data will be computed numerically and analysed in the Clermont-Ferrand center. A descriptive analysis will be proposed as the expected number of patients affected by this rare disease varies from 10 to 30. Median []interquartiles], means [standard deviation] and percentages will be calculated for quantitative data.

Collected data will include :

* general information :

  * centre number
  * Patient (First letter last name, first letter first name)
  * Investigator name
  * Patient age
  * Patient sex
  * Age at clinical onset
  * Patient alive or deceased
  * Age when deceased
  * Ethnic origin
  * Consanguinity
* Clinical data :

  * Birth term
  * Age at sitting
  * Age at walking
  * Age at first language
  * Acquisition of fine motor skills
  * Autistic troubles
  * motor regression and age
  * Loss of walking and age
  * Language regression and age
  * Social skill regression and age
  * Vision loss and age
  * Hearing loss and age
  * Progressivity of symptoms
  * Axial hypotonia
  * Ataxia
  * Dystonia
  * Parkinsonism
  * Other paroxysmic movements
  * Spasticity
  * Hyperreflexia
  * Hyporeflexia /areflexia
  * Babinski sign
  * Peripheral neuropathy
  * Muscular atrophy
  * Bulbar signs
  * Dysarthria
  * Nystagmus
  * Strabism
  * Seizures
  * Intellectual deficiency and severity
  * Specific learning disabilities
  * Behavioral troubles
  * Mood disorders
  * Scoliosis
  * Other orthopedic abnormalities
  * Sleep disturbance or Sleep apnea syndrome
  * Gastro-intestinal troubles
  * Other symptoms
  * Patient still ambulant or not
  * Gross Motor Function Classification Score (GMFCS from 1 to 5)
  * Schooling modalities
  * Eye fundus abnormalities
* Genetic data :

  - Name of mutation 1 / mutation 2 in PLA2G6
* Radiological data :

  * Iron deposits
  * White matter abnormalities
  * Cerebellar atrophy
  * Optic nerve atrophy
  * Brainstem atrophy
  * Cortical-subcortical atrophy
  * Splenium verticalization
  * Other abnormalities of corpus callosum
  * Clava hypertrophy
  * Other abnormalities
* Electrophysiological data :

  * abnormalities of EEG
  * abnormalities of electromyogram
  * Other results of evoked potentials
* Pathophysiological data:

  * Results of potential cutaneous, muscular, nervous or other biopsies
  * Results of potential autopsy in case of deceased patients
* Therapeutical data :

  * Type of feeding (oral, tube..)
  * Ventilatory support
  * Baclofen
  * Botulinic toxin
  * L-dopa
  * Trihexyphenidyl
  * Tetrabenazine
  * Antiepileptic drugs (names)
  * neuropathic analgesic
  * Treatment os swallowing
  * Mitochondrial cocktail or other vitamins
  * Treatment of sleep disorders
  * Orthopedic or other surgery
  * Other symptomatic treatment
  * Treatment leading to aggravation
  * Treatment leading to improvement

ELIGIBILITY:
Inclusion Criteria:

* Children with atypical neuroaxonal dystrophy under 18 years at disease-onset
* with 2 deleterious mutations in the PLA2G6 gene
* alive or deceased
* Non-opposition of parents to participate to the retrospective study

Exclusion Criteria:

* Classical form of infantile neuroaxonal dystrophy
* Neuro-axonal dystrophy with adult-onset
* Opposition of parents to participate to the retrospective study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will be recruited from a French retrospective cohort on invitation to neuropaeditricians exercing in French pediatric hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Birth term in gestational weeks | through study completion, an average of 9 months
  quantitative feature, number of gestational weeks
Age at sitting in months | through study completion, an average of 9 months
  quantitative feature, age in months
Age at walking in years and months | through study completion, an average of 9 months
  quantitative feature, age in years and months
Age at first language in years and months | through study completion, an average of 9 months
  quantitative feature, age in years and months
Acquisition of fine motor skills | through study completion, an average of 9 months
  Qualitative feature, answer :Yes / No
Autistic troubles | through study completion, an average of 9 months
  Qualitative feature, answer :Yes / No
Neurological regression | through study completion, an average of 9 months
  Qualitative feature, answer :Yes / No Precision of age at onset Precision of type of regression (language, motor, social, hearing, visual)
Progressivity of symptoms | through study completion, an average of 9 months
  Qualitative feature, answer :Yes / No
Axial hypotonia | through study completion, an average of 9 months
  Qualitative feature, answer :Yes / No
Movement disorders | through study completion, an average of 9 months
  Qualitative feature, answer :Yes / No Precision of age at onset Precision of type (dystonia, paroxysmal dyskinesia, parkinsonism, nystagmus, ataxia, other)
Pyramidal signs | through study completion, an average of 9 months
  Qualitative feature, answer :Yes / No Precision of age at onset Precision of type (spasticity, Babinski, hyperreflexia, other)
Intellectual deficiency | through study completion, an average of 9 months
  Qualitative feature, answer :Yes / No Precision of severity (mild, moderate, severe, profound)
Peripheral neurological signs | through study completion, an average of 9 months
  Qualitative feature, answer :Yes / No Precision of age at onset Precision of type (myopathy, neuropathy, areflexia, bulbar signs, other)
Seizures | through study completion, an average of 9 months
  Qualitative feature, answer :Yes / No Precision of age at onset
Behavioral or mood disorders | through study completion, an average of 9 months
  Qualitative feature, answer :Yes / No Precision of age at onset Precision of type
Orthopaedic disorders | through study completion, an average of 9 months
  Qualitative feature, answer :Yes / No Precision of age at onset Precision of type (scoliosis, hip, ankle deformations, other)
Sleep disorders | through study completion, an average of 9 months
  Qualitative feature, answer :Yes / No Precision of age at onset Precision of type
Gastro-intestinal disorders | through study completion, an average of 9 months
  Qualitative feature, answer :Yes / No Precision of age at onset Precision of type
Visual abnormalities | through study completion, an average of 9 months
  Qualitative feature, answer :Yes / No Precision of age at onset Precision of type (strabism, nystagmus, eye fundus abnormalities, other)
Radiological abnormalities | through study completion, an average of 9 months
  Qualitative feature, answer :Yes / No Precision of age at onset Precision of type (Iron deposits, White matter abnormalities, Cerebellar atrophy, Optic nerve atrophy, Brainstem atrophy, Cortical-subcortical atrophy, Splenium verticalization, Other abnormalities of corpus callosum, Clava hypertrophy, Other)
GMFCS | through study completion, an average of 9 months
  GMFCS scoring from 1 to 5

SECONDARY OUTCOMES:
Mutations in PLA2G6 | through study completion, an average of 9 months
  Qualitative feature, answer Yes / No Precision of the name of mutation 1 / name of mutation 2 in the PLA2G6 gene for each patient
Electrophysiological findings | through study completion, an average of 9 months
  Qualitative feature, answer : Yes / No Precision of type (abnormalities of EEG, abnormalities of electromyogram, abnormalities of evoked potentials)
Pathophysiological findings | through study completion, an average of 9 months
  Qualitative feature, answer : Yes / No Precision of type (abnormalities on cutaneous, muscular, nervous or other biopsies abnormalities on autopsy)
Therapeutics | through study completion, an average of 9 months
  Qualitative feature, answer Yes / No Precision of type and age at onset (feeding tube / Ventilatory support / Baclofen / Botulinic toxin/ L-dopa/ Trihexyphenidyl/ Tetrabenazine / Antiepileptic drugs / Neuropathic analgesic / Treatment of swallowing / Mitochondrial cocktail or other vitamins / Treatment of sleep disorders / Orthopedic or other surgery / Other) Precision of aggravation / improvement
Phenotype-genotype correlation | through study completion, an average of 9 months
  Secondary analysis of phenotype-genotype correlation

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Sarret, Study Director — University Hospital, Clermont-Ferrand
Locations (7):
- France (7):
  - CHU clermont-ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - HCL, Hôpital Femme, mère, enfant, Lyon
  - CHU Montpellier, Montpellier
  - APHP, Paris
  - CHU Rennes, Rennes
  - CHU Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davids M, Kane MS, He M, Wolfe LA, Li X, Raihan MA, Chao KR, Bone WP, Boerkoel CF, Gahl WA, Toro C. Disruption of Golgi morphology and altered protein glycosylation in PLA2G6-associated neurodegeneration. J Med Genet. 2016 Mar;53(3):180-9. doi: 10.1136/jmedgenet-2015-103338. Epub 2015 Dec 14. PMID 26668131
- [Background] Erro R, Balint B, Kurian MA, Brugger F, Picillo M, Barone P, Bhatia KP, Pellecchia MT. Early Ataxia and Subsequent Parkinsonism: PLA2G6 Mutations Cause a Continuum Rather Than Three Discrete Phenotypes. Mov Disord Clin Pract. 2016 Mar 31;4(1):125-128. doi: 10.1002/mdc3.12319. eCollection 2017 Jan-Feb. PMID 30868093
- [Background] Yamashita C, Funayama M, Li Y, Yoshino H, Yamada H, Seino Y, Tomiyama H, Hattori N. Mutation screening of PLA2G6 in Japanese patients with early onset dystonia-parkinsonism. J Neural Transm (Vienna). 2017 Apr;124(4):431-435. doi: 10.1007/s00702-016-1658-7. Epub 2016 Dec 9. PMID 27942883
- [Background] Shi CH, Tang BS, Wang L, Lv ZY, Wang J, Luo LZ, Shen L, Jiang H, Yan XX, Pan Q, Xia K, Guo JF. PLA2G6 gene mutation in autosomal recessive early-onset parkinsonism in a Chinese cohort. Neurology. 2011 Jul 5;77(1):75-81. doi: 10.1212/WNL.0b013e318221acd3. Epub 2011 Jun 22. PMID 21700586
- [Background] Yoshino H, Tomiyama H, Tachibana N, Ogaki K, Li Y, Funayama M, Hashimoto T, Takashima S, Hattori N. Phenotypic spectrum of patients with PLA2G6 mutation and PARK14-linked parkinsonism. Neurology. 2010 Oct 12;75(15):1356-61. doi: 10.1212/WNL.0b013e3181f73649. PMID 20938027
- [Background] Paisan-Ruiz C, Bhatia KP, Li A, Hernandez D, Davis M, Wood NW, Hardy J, Houlden H, Singleton A, Schneider SA. Characterization of PLA2G6 as a locus for dystonia-parkinsonism. Ann Neurol. 2009 Jan;65(1):19-23. doi: 10.1002/ana.21415. PMID 18570303
- [Background] McMillan HJ, Marshall AE, Venkateswaran S, Hartley T, Warman-Chardon J, Ramani AK, Marshall CR, Michaud J, Boycott KM, Dyment DA, Kernohan KD. Whole genome sequencing reveals biallelic PLA2G6 mutations in siblings with cerebellar atrophy and cap myopathy. Clin Genet. 2021 May;99(5):746-748. doi: 10.1111/cge.13935. Epub 2021 Feb 11. No abstract available. PMID 33576074
- [Background] Koh K, Ichinose Y, Ishiura H, Nan H, Mitsui J, Takahashi J, Sato W, Itoh Y, Hoshino K, Tsuji S, Takiyama Y; Japan Spastic Paraplegia Research Consotium. PLA2G6-associated neurodegeneration presenting as a complicated form of hereditary spastic paraplegia. J Hum Genet. 2019 Jan;64(1):55-59. doi: 10.1038/s10038-018-0519-7. Epub 2018 Oct 9. PMID 30302010
- [Background] Ozes B, Karagoz N, Schule R, Rebelo A, Sobrido MJ, Harmuth F, Synofzik M, Pascual SIP, Colak M, Ciftci-Kavaklioglu B, Kara B, Ordonez-Ugalde A, Quintans B, Gonzalez MA, Soysal A, Zuchner S, Battaloglu E. PLA2G6 mutations associated with a continuous clinical spectrum from neuroaxonal dystrophy to hereditary spastic paraplegia. Clin Genet. 2017 Nov;92(5):534-539. doi: 10.1111/cge.13008. Epub 2017 Apr 19. PMID 28295203
- [Background] Jain S, Bhasin H, Romani M, Valente EM, Sharma S. Atypical Childhood-onset Neuroaxonal Dystrophy in an Indian Girl. J Pediatr Neurosci. 2019 Apr-Jun;14(2):90-93. doi: 10.4103/jpn.JPN_91_18. PMID 31516627
- [Background] Salih MA, Mundwiller E, Khan AO, AlDrees A, Elmalik SA, Hassan HH, Al-Owain M, Alkhalidi HM, Katona I, Kabiraj MM, Chrast R, Kentab AY, Alzaidan H, Rodenburg RJ, Bosley TM, Weis J, Koenig M, Stevanin G, Azzedine H. New findings in a global approach to dissect the whole phenotype of PLA2G6 gene mutations. PLoS One. 2013 Oct 9;8(10):e76831. doi: 10.1371/journal.pone.0076831. eCollection 2013. PMID 24130795
- [Background] Gregory A, Kurian MA, Maher ER, Hogarth P, Hayflick SJ. PLA2G6-Associated Neurodegeneration. 2008 Jun 19 [updated 2017 Mar 23]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1675/ PMID 20301718
- [Background] Romani M, Kraoua I, Micalizzi A, Klaa H, Benrhouma H, Drissi C, Turki I, Castellana S, Mazza T, Valente EM, Gouider-Khouja N. Infantile and childhood onset PLA2G6-associated neurodegeneration in a large North African cohort. Eur J Neurol. 2015 Jan;22(1):178-86. doi: 10.1111/ene.12552. Epub 2014 Aug 27. PMID 25164370
- [Background] Kurian MA, Hayflick SJ. Pantothenate kinase-associated neurodegeneration (PKAN) and PLA2G6-associated neurodegeneration (PLAN): review of two major neurodegeneration with brain iron accumulation (NBIA) phenotypes. Int Rev Neurobiol. 2013;110:49-71. doi: 10.1016/B978-0-12-410502-7.00003-X. PMID 24209433
- [Background] Illingworth MA, Meyer E, Chong WK, Manzur AY, Carr LJ, Younis R, Hardy C, McDonald F, Childs AM, Stewart B, Warren D, Kneen R, King MD, Hayflick SJ, Kurian MA. PLA2G6-associated neurodegeneration (PLAN): further expansion of the clinical, radiological and mutation spectrum associated with infantile and atypical childhood-onset disease. Mol Genet Metab. 2014 Jun;112(2):183-9. doi: 10.1016/j.ymgme.2014.03.008. Epub 2014 Mar 29. PMID 24745848
- [Background] Gregory A, Polster BJ, Hayflick SJ. Clinical and genetic delineation of neurodegeneration with brain iron accumulation. J Med Genet. 2009 Feb;46(2):73-80. doi: 10.1136/jmg.2008.061929. Epub 2008 Nov 3. PMID 18981035
- [Background] Kurian MA, Morgan NV, MacPherson L, Foster K, Peake D, Gupta R, Philip SG, Hendriksz C, Morton JE, Kingston HM, Rosser EM, Wassmer E, Gissen P, Maher ER. Phenotypic spectrum of neurodegeneration associated with mutations in the PLA2G6 gene (PLAN). Neurology. 2008 Apr 29;70(18):1623-9. doi: 10.1212/01.wnl.0000310986.48286.8e. PMID 18443314
- [Background] Khateeb S, Flusser H, Ofir R, Shelef I, Narkis G, Vardi G, Shorer Z, Levy R, Galil A, Elbedour K, Birk OS. PLA2G6 mutation underlies infantile neuroaxonal dystrophy. Am J Hum Genet. 2006 Nov;79(5):942-8. doi: 10.1086/508572. Epub 2006 Sep 19. PMID 17033970
- [Background] Morgan NV, Westaway SK, Morton JE, Gregory A, Gissen P, Sonek S, Cangul H, Coryell J, Canham N, Nardocci N, Zorzi G, Pasha S, Rodriguez D, Desguerre I, Mubaidin A, Bertini E, Trembath RC, Simonati A, Schanen C, Johnson CA, Levinson B, Woods CG, Wilmot B, Kramer P, Gitschier J, Maher ER, Hayflick SJ. PLA2G6, encoding a phospholipase A2, is mutated in neurodegenerative disorders with high brain iron. Nat Genet. 2006 Jul;38(7):752-4. doi: 10.1038/ng1826. Epub 2006 Jun 18. PMID 16783378